CLINICAL TRIAL: NCT04421144
Title: Accuracy of CAD/CAM Cutting Guides and Customized Titanium Plates for Virtual Planning Transfer in Bimaxillary Orthognathic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Zain, assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dr.Zain protocol
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Evaluation of the Accuracy of Transferring the Virtual Planning to the Surgery
Keywords: CAD/CAM; orthognathic surgery; virtual planning; cutting guides; customized titanium plates
MeSH Terms: interventions — Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): using CAD/CAM surgical cutting guides for maxilla and mandible and customized titanium plates to guide all osteotomies and fixation of both arches.
  Interventions: Procedure: orthognathic surgery

INTERVENTIONS:
Procedure: orthognathic surgery — patients with maxillofacial disharmony will undergo orthognathic surgery using CAD/CAM Cutting Guides and Customized Titanium Plates.

SUMMARY:
In this research, we aim to use CAD/CAM surgical cutting guides for maxilla and mandible and customized titanium plates to guide all osteotomies and fixation of both arches.

DETAILED DESCRIPTION:
Intervention:

1. Diagnostic procedure:

   All Patients will be selected according to inclusion and exclusion criteria & Comprehensive clinical examination and understanding of patients' chief complains and needs will be carried out.

   Preoperative patient photographs (Frontal, Profile, 45°, smile, and dental occlusion).

   Alginate Impressions of upper & lower jaws will be taken for acquiring diagnostic dental casts.

   A heat-cured acrylic resin stent will be constructed on the stone model. Using the stent, a radiographic stent will be constructed for imaging and planning procedures.

   Cone Beam Computed Topography (CBCT) for the patients will be carried out. All patients will be referred to an orthodontist for presurgical phase of orthodontic treatment for decompensation and to attain stable occlusion in three points in the surgery.
2. Planning procedure:

   All planning procedures are carried out by MZ and under the supervision of AH and MH.

   Computer-aided planning & MCROS design for all patients: All planning will be done using specialized software .

   One virtual 3D anatomic model of the patient will be constructed through thresholding & image fusion.

   Virtual Le Fort I osteotomy and then the maxilla will be virtually adjusted according to the facial symmetry planes and clinical anthropometric analysis. Virtual simulation of the sagittal split of the mandible will be performed and the mandible position adjusted according to the bite registered.

   After settling on the optimum virtual plan, designing of the cutting guides and titanium plates will then be started.
3. Intra-operative procedures:

   The surgical procedures will be carried out by MZ under the supervisor of AH in the Oral & Maxillofacial operating floor on the 8th floor of the faculty of Oral & Dental Medicine new building.

   Scrubbing and draping of the patient will be carried out in a standard fashion according to Anon 2006.

   Local anaesthesia (lidocaine 2%, 1/100000 adrenaline) will be injected intraorally along the incision lines for hemostasis.

   Access through a vestibular intraoral incision for maxilla & Sagittal split incision for mandible will be carried out. Dissection and reflection to reach the bone will be carried out.

   Le Fort I Maxillary & Bilateral Sagittal split mandibular osteotomies will be carried out using the osteotomy cutting guides.

   Complete mobilization of maxillary and mandibular segments. Reposition and fixation of the maxillary & mandibular segments using customized titanium plates.

   The incisions will be closed with continuous mattress resorbable sutures .
4. Post-operative care:

   Patients will start antibiotics 4 hours after the last intraoperative dose (Amoxicillin / Clavulanic acid 625 mg every 8 hours) for 5 days Patients will start analgesics (NSAIDs every 6 hours) for 3 days Mouthwash (Chlorhexidine 0.12%) will be prescribed for 2 more weeks.
5. Criteria for discontinuing or modifying intervention:

   * Difficulty with the use of cutting guides and customized titanium plates.
   * Inaccurate translation of the surgical plan.
6. Strategies to improve adherence to intervention:

   Postoperative orthodontic treatment is necessary after the operation to obtain the final stable occlusion.
7. Concomitant care:

   Not needed.
8. Follow up & Evaluation:

Post-operative treatment will start immediately postoperative (4 hours). The patients will be scheduled for follow-up visits weekly for a month then on a monthly basis for 5 more months.

Within the first week postoperatively CBCT using same parameters will be ordered to calculate the difference between surgical plan and actual outcome will be evaluated.

Patient will be referred back to the orthodontist to receive his postsurgical orthodontics 4-6 weeks postoperatively.

The technique will be evaluated by applying hard tissue parameters to compare the virtual orthognathic planning (P0) with the postoperative result (P1) using 3D cephalometry and image fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dentofacial disharmony and misalignment requiring bimaxillary orthognathic surgeries.
2. Patients with no signs or symptoms of active TMDs.
3. Highly motivated patients.

Exclusion Criteria:

1. Patients who refused to be included in the research.
2. Patients with systemic diseases that may hinder the normal healing process or render the patient not fitting for general anaesthesia.
3. Patients with intra-bony lesions or infections that may retard the osteotomy healing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the surgical transfer | within first week postoperatively
  Computer software on pre/postoperative CBCT

SECONDARY OUTCOMES:
Patient satisfaction: Visual analog scale (questionnaire) | one week postoperative
  Visual analog scale (questionnaire)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol